CLINICAL TRIAL: NCT06856876
Title: Examining the Effectiveness of Multidisciplinary Care Teams in Improving Outcomes for Breast Cancer Patients
Acronym: MDCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yousaf Jan (Other Government)
Responsible Party: Sponsor-Investigator, Yousaf Jan, Principal investigator, Hayat Abad Medical Complex, Peshawar
Organization: Hayat Abad Medical Complex, Peshawar (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMCKP2
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancers; Breast Cancer Female; Breast Cancer Stage I
Keywords: Breast Cancer; MDCT; Disease free survival; Quality of life; outcome
MeSH Terms: conditions — Breast Neoplasms | interventions — Patient Care Team; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDCT (Group A) (Experimental): Participants receive multidisciplinary care team (MDCT) treatment, including personalized treatment plans developed by oncologists, radiologists, and surgeons.
  Interventions: Other: Multidisciplinary Care Team (MDCT) Approach
- Standard Therapy (Group B) (Active Comparator): Participants receive standard care for breast cancer according to the current institutional protocols.
  Interventions: Other: Standard Breast Cancer Therapy

INTERVENTIONS:
Other: Multidisciplinary Care Team (MDCT) Approach — A personalized breast cancer treatment plan developed through regular case discussions by a team of radiologists, oncologists, and surgeons. The MDCT coordinates patient support services and tracks treatment progress according to evidence-based guidelines.
  Other Names: MDCT
  Arms: MDCT (Group A)
Other: Standard Breast Cancer Therapy — Breast cancer treatment provided according to the institutional protocols at Hayatabad Medical Complex, including standard surgery, chemotherapy, and/or radiotherapy as clinically indicated.
  Other Names: Standard Therapy
  Arms: Standard Therapy (Group B)

SUMMARY:
To compare clinical outcomes, patient-reported measures (PROMs), and healthcare utilization between standard care with or without an MDCT in a cohort of women treated for breast cancer.

DETAILED DESCRIPTION:
This single-center, prospective interventional trial evaluates the effectiveness of Multidisciplinary Care Teams (MDCTs) in improving outcomes for newly diagnosed breast cancer patients at Hayatabad Medical Complex, Peshawar. The study enrolled 73 participants from May 2021 to April 2024, with follow-up sessions every six months for up to two years.

Participants were randomly assigned to two groups:

Group A (n=37): Received care through MDCTs, which included radiologists, oncologists, and surgeons collaborating to create personalized treatment plans and monitor patient progress.

Group B (n=36): Received standard therapy according to existing institutional protocols.

The study assesses multiple outcomes, including **disease-free survival (DFS), overall survival (OS), recurrence rates, complication rates, patient-reported outcomes (PROs), quality of life (measured via SF-36), and healthcare utilization.

Statistical analyses include Kaplan-Meier survival curves, log-rank tests, Cox proportional hazards regression models, repeated-measures ANOVA, and linear regression models to identify predictors of survival and quality of life.

The study protocol was approved by the Institutional Review Board (IRB) and complies with the Declaration of Helsinki. All participants provided informed consent prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

All female patients, diagnosed with breast cancer

Exclusion Criteria:

Previous treatment for breast cancer, concurrent enrollment in another clinical research, and serious medical conditions that could affect study outcomes

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biologically female patients diagnosed with breast cancer are eligible to participate
Enrollment: 73 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | 24 months (measured at 6, 12, 18, and 24 months)
  Time from the start of treatment to the first occurrence of disease relapse, progression, or death from any cause.
Overall survival | 24 months (measured at 6, 12, 18, and 24 months)
  Time from the start of treatment until death from any cause.

SECONDARY OUTCOMES:
Recurrence rate | 24 months (measured at 6, 12, 18, and 24 months)
  Number of participants with local or distant breast cancer recurrence.
Complication rate | 24 months (measured at 6, 12, 18, and 24 months)
  Incidence of treatment-related complications (e.g., surgical site infections, chemotherapy side effects).

CONTACTS AND LOCATIONS:
Overall Officials: Yousaf Jan, MBBS, FCPS, FRCS, MRCS, ECFMG, Principal Investigator — Hayat Abad Medical Complex, Peshawar
Locations (1):
- Hayatabad Medical Complex, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) due to confidentiality concerns and institutional policies.